CLINICAL TRIAL: NCT04712201
Title: En Bloc Bladder Tumor Resection: Prospective Randomized Evaluation of Monopolar, Bipolar and Laser Energy
Brief Title: En Bloc Bladder Tumor Resection: Prospective Randomized Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Puigvert (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Principal Investigator, Alberto Breda, Chief of the Uro-Oncology Division and Kidney Transplant Unit, Fundacio Puigvert
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017/09c
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Urothelial Carcinoma Bladder; Bladder Cancer
Keywords: TURBT; En bloc; Urothelial cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- En bloc (Experimental): En bloc transurethral resection of the bladder
  Interventions: Procedure: En bloc transurethral resection of bladder tumor (TURBT)
- Conventional (Active Comparator): Conventional transurethral resection of the bladder
  Interventions: Procedure: Conventional TURBT

INTERVENTIONS:
Procedure: En bloc transurethral resection of bladder tumor (TURBT) — En bloc transurethral resection of bladder tumor using thulium:yttrium aluminium garnet, monopolar and bipolar energy
  Arms: En bloc
Procedure: Conventional TURBT — Conventional transurethral resection of bladder tumor using monopolar and bipolar energy
  Arms: Conventional

SUMMARY:
INTRODUCTION Bladder tumor is the second most common neoplasm in the genitourinary tract. Most cases of ex novo diagnosis of bladder cancers are present as non-invasive muscle tumors, which are treatable through endourological procedures. The current standard is based on conventional transurethral resection of bladder tumor, although high rates of recurrence have been reported following resection of the primary tumor. Given the importance of a correct initial diagnosis in these cases, en bloc transurethral resection has developed over the past 2 decades. This technique was born, according to the literature, with 3 main objectives: to improve the quality of the surgical piece for its anatomopathological reading, reduce the rate of postoperative complications and reduce the rate of relapses in the surgical bed. This technique is used as a common practice of tumor resection in other centers and has been shown in multiple publications that it does not increase surgical risk or negatively affect cancer results.

OBJECTIVE The objective of our study is to compare feasibility, perioperative complication rate, accuracy of staging and recurrence/progression rates when performing en bloc resection by means of different energies: monopolar, bipolar and laser energy.

MATERIAL AND METHODS Between April 2018 and June 2021, a prospective randomized study will be conducted including patients undergoing a transurethral resection of initial or recurrent bladder tumor, either unifocal or multifocal. Patients with tumors less than 3 cm and with less than 3 tumors shall be included if multiple. Patients with more than 3 tumors or tumors over 3cm, those with evidence of invasive muscle tumor(cT2) or those with evidence of remote metastasis, whether lymphatic or organic, will be excluded.

Patients will be randomized into two groups:

* Group 1 (test): en bloc resection (n-180). It will be divided into 3 subgroups according to the energy used (monopolar, bipolar, laser energy).
* Group 2 (control): Conventional transurethral resection (n-120). It will be divided into 2 subgroups depending on the energy used (monopolar or bipolar).

A fact sheet will be given to the patient about the study and the signature of the informed consent will be requested in order to be included. The patient will be free to leave the study at any time without having to provide any justification and without affecting the treatment, intervention and follow-up that must be carried out.

The processing and storage of samples will be carried out in the pathological anatomy laboratory, according to standard clinical practice.

Patients will be monitored according to the usual clinical practice protocol (minimum 5-year follow-up), included in the non-muscle invasive bladder tumor protocols of the Puigvert Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Unifocal primary or recurrent bladder cancer with size less or equal than 3 cm
* Multifocal primary or recurrent bladder cancer less or equal than 3 lesions and with size less or equal than 3 cm

Exclusion Criteria:

* Evidence of > 3 tumors or > 3 cm
* Computed tomography/cystoscopy suspect of muscle-invasive bladder cancer (cT2 or higher)
* Computed tomography/magnetic resonance evidence of distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Staging of bladder tumor | Three years
  Evaluation of muscle presence in the specimen

SECONDARY OUTCOMES:
Intraoperative complications | Three years
  Bladder perforation grading, obturatory reflex, conversions to conventional TURB
Rate of planned adjuvant treatment | Three years
  Rate of planned postoperative single instillation of mitomycin/epirubicin
Post-operative complications | Three years
  Post-operative complications according to Clavien-Dindo System
Substaging T1 bladder cancer | Three years
  T1a, T1b and T1c
Recurrence-free survival | Through study completion, an average of five years
  Recurrence of bladder cancer
Progression-free survival | Through study completion, an average of five years
  Progression of bladder cancer
Disease-free survival | Through study completion, an average of five years
  Disease-free survival
Cancer specific survival | Through study completion, an average of five years
  Cancer specific survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacio Puigvert, Barcelona, Spain

REFERENCES:
- [Derived] Gallioli A, Diana P, Fontana M, Territo A, Rodriguez-Faba O, Gaya JM, Sanguedolce F, Huguet J, Mercade A, Piana A, Aumatell J, Bravo-Balado A, Algaba F, Palou J, Breda A. En Bloc Versus Conventional Transurethral Resection of Bladder Tumors: A Single-center Prospective Randomized Noninferiority Trial. Eur Urol Oncol. 2022 Aug;5(4):440-448. doi: 10.1016/j.euo.2022.05.001. Epub 2022 May 23. PMID 35618567